CLINICAL TRIAL: NCT03607071
Title: Outcome of Myocardial Inflammation After Steroid Therapy in Thai Systemic Sclerosis Patients: an Open Label Study
Brief Title: Outcome of Steroid Therapy for Myocardial Inflammation in Scleroderma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Chingching Foocharoen, Principle investigator, Khon Kaen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSc-KKU
Record Dates: First submitted 2018-07-20; First posted 2018-07-31 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Myocardial Inflammation
MeSH Terms: conditions — Myocarditis | interventions — Prednisolone

STUDY DESIGN:
Intervention Model Description: Moderate dose steroid therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prednisolone (Experimental): The patient who has detected myocardial inflammation from cardiac MRI from baseline is given prednisolone 30 mg/d and taper 5-10 mg per 2 weeks until off at week 24.
  Interventions: Drug: Prednisolone and taper

INTERVENTIONS:
Drug: Prednisolone and taper — Prednisolone 30 mg/d and taper 5-10 mg per 2 weeks until off at week 24.
  Other Names: Moderate steroid therapy

SUMMARY:
Primary myocardial involvement is common in scleroderma, effected to pericardium, vascular, conducting defect and especially myocardium. Cardiac MRI is widely used for assessment of cardiac involvement in scleroderma, both structural and functional pathology. Cardiac MRI has a diagnostic accuracy of 85% for the detection of myocardial inflammation. Nowadays, the treatment of myocardial inflammation in scleroderma is uncertain. The investigator's study aims to define the cardiac outcome after moderate dose steroid therapy in the patients who have myocardial inflammation detection by cardiac MRI.

ELIGIBILITY:
Inclusion Criteria:

• The adult scleroderma patients who were defined as having myocardial inflammation by cardiac MRI.

Exclusion Criteria:

* Current infection that needs systemic antibiotic therapy
* Active viral hepatitis B or C
* Uncontrolled diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Changing of degree of myocarditis evaluated by cardiac MRI after treatment compare to baseline | 24 weeks
  Myocarditis is defined as inflammatory disease of the myocardium according to the cardiac MRI Lake Louise criteria at least 2 of the following criteria:
  1. Regional or global myocardial signal intensity increased in the T2-weighted images;
  2. Increased global myocardial early enhancement ratio between the myocardium and skeletal muscle in the gadolinium-enhanced T1-weighted images; and,
  3. At least 1 focal lesion with nonischemic regional distribution in the inversion-recovery-prepared, gadolinium-enhanced, T1-weighted images (delayed enhancement).
  Response to treatment is defined as any reducing of degree of myocarditis without any progression of myocardial fibrosis or scarring when compared to the cardiac MRI baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine, Faculty of Medicine, Khon Kaen University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pussadhamma B, Tipparot T, Chaosuwannakit N, Mahakkanukrauh A, Suwannaroj S, Nanagara R, Foocharoen C. Clinical Outcomes of Myocarditis after Moderate-Dose Steroid Therapy in Systemic Sclerosis: A Pilot Study. Int J Rheumatol. 2020 Dec 19;2020:8884442. doi: 10.1155/2020/8884442. eCollection 2020. PMID 33414828